CLINICAL TRIAL: NCT05638776
Title: A Multicenter, Randomized, Single-Blind, Placebo-Parallel-Controlled Research of REGEND001 Cell Therapy for Treatment of Chronic Obstructive Pulmonary Disease (COPD) With Diffusion Capacity Defect
Brief Title: Treatment of Chronic Obstructive Pulmonary Disease (COPD) With Diffusion Capacity Defect by REGEND001 Cell Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Southwest Hospital, China (Other); Shanghai Zhongshan Hospital (Other); China-Japan Friendship Hospital (Other); Shanghai East Hospital (Other); Regend Therapeutics XLotus (Jiangxi) Co, Ltd. (Unknown); The First Affiliated Hospital of Nanchang University (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGEND001-COPD-201
Record Dates: First submitted 2022-11-02; First posted 2022-12-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REGEND001 cell therapy (Experimental): REGEND001 cell therapy
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGEND001 cell therapy — Transplantation of the cell product
Drug: Placebo — Transplantation of Placebo
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the third leading cause of death worldwide with the characterization of obstructed airflow. In a large number of patients, diffusion function is impaired along with the progression of disease. REGEND001 cell therapy, comprised of airway basal cells with ability to regenerate lung tissue, is promising to COPD treatment. In this study, a multicenter, randomized, single-blind, placebo-parallel-controlled trial is performed to assess the efficacy and safety of REGEND001 cell therapy in treatment of chronic obstructive pulmonary disease with diffusion capacity defect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 40 to 75 at the time of signing informed consent.
* Diagnosed with COPD according to the 2021 Global Initiative for Chronic Obstructive Lung Disease (GOLD).
* The ratio of forced expiratory volume in one second (FEV1)/forced vital capacity (FVC)FEV1/FVC is < 70% after inhalation of bronchodilators.
* The diffusion function of carbon monoxide (DLCO) is ≥ 20% and < 80% of the predicted value at screening.
* Tolerated to pulmonary function tests.
* Tolerated to bronchoscopy
* Voluntary to sign the informed consent, coordinated to finish the trial-related procedures and tests, and capable of recording or stating the change of disease condition in a relatively complete manner.

Exclusion Criteria:

* Females who are pregnant, nursing, or planning to be pregnant within a year after using this product (or males whose spouse planning to be pregnant);
* Subject positive in each of the tests containing treponema pallidum antibody (TP-Ab), human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody at screening. But except the followings:

  1. Hepatitis B virus carriers (only HBsAg positive without any hepatitis symptom or sign, and all liver function tests present normal results or abnormal markers without clinical significance by the assessment of investigators);
  2. Cured hepatitis C patients (negative in HCV ribonucleic acid (RNA) test);
* Subject with assessed survival time of < 1 year by investigators at screening;
* Subject with malignant tumors or a history of malignant tumors at screening;
* Subject with infections in lung or other sites, requiring intravenous drug treatment within a week prior to screening;
* Subject with more than 4 moderate-to-severe AECOPD, resulting in hospitalization within a year prior to screening;
* Subject with one or more pathogenetic or serologic findings of the novel coronavirus infection, or symptoms of suspected infection within 6 weeks prior to screening;
* Subject with a history of invasive or noninvasive mechanical ventilation within 4 weeks prior to screening;
* Subject who has taken prednisone tablets orally at a dose of ≥ 20 mg/day (or equivalent amount of other oral corticosteroids) within 4 weeks prior to screening;
* Subject with major lung diseases other than COPD by assessment of investigators at screening;
* Subject with severe systemic diseases other than lung within 6 months prior to screening and assessed to be inappropriate to participate in this trial by investigators;
* Subject with severe anemia or poorly controlled granulocyte deficiency, thrombocytopenia by assessment of investigators;
* Subject with abnormal coagulation and assessed to be negative for the safety of fiberoptic bronchoscopy operations at screening;
* Subject requiring long-term anticoagulation therapy of using antiplatelet coagulant therapeutic agents and disable to discontinue their medications 1 week prior to cell collection and cell infusion as assessed by investigators;
* Subject with a risk of suicide, a history of mental illness or a history of epilepsy at screening;
* Subject with severe arrhythmias or heart conduction disorders (degree II or above) in 12-lead ECG test at screening;
* Subject participated in other clinical trials with interventions within 3 months prior to screening;
* Investigators, co-investigators, research coordinators, employees of research participants or research centers, or their family members;
* Any circumstance considered to probably increase the risk of patients or interfere with the clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Change of lung diffusing capacity for carbon monoxide (DLCO) from baseline | Within 52 weeks after treatment
  DLCO is considered a measure of the conductance of CO across the alveolar-capillary membrane and its binding with hemoglobin.

SECONDARY OUTCOMES:
Change of the alveolar volume (VA) from baseline | Winthin 52 weeks after treatment
  Alveolar ventilation is the exchange of gas between the alveoli and the external environment. It is the process by which oxygen is brought into the lungs from the atmosphere and by which the carbon dioxide carried into the lungs in the mixed venous blood is expelled from the body.
Change of images of lung by high resolution computed tomography (HR-CT) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  HR-CT images of lung will be analyzed to indicate the change of pulmonary structure.
Change of forced vital capacity (FVC) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  FVC is the full amount of air that can be exhaled with effort in a complete breath.
Change of forced expiratory volume in one second (FEV1) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  FEV1 is the volume of breath exhaled with effort in one second.
Change of forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  The FEV1/FVC is a ratio that reflects the amount of air you can forcefully exhale from your lungs. It's measured by spirometry, a test used to evaluate lung function.
Change of the diffusing capacity for carbon monoxide/ the alveolar volume (DLCO/VA) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  The DLCO test refers to the diffusing capacity for carbon monoxide in the lungs. It's a type of pulmonary function test that helps to assess how well gas is exchanged between the lungs and the bloodstream.Since DLCO is affected by the amount of inhaled gas and lung volume, the subject's alveolar ventilation (VA) is also considered when evaluating diffusion function to exclude the effect of lung volume on diffusion volume.
Change of 6-minute-walk test (6MWT) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  The 6MWT is a commonly used test for the objective assessment of functional exercise capacity by testing the distance patients can walk at the fastest speed within 6 minutes.
Change of modified medical research council (mMRC) dyspnea scale from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  It is a questionnaire to evaluate how breathlessness impacts daily activities. According to the degree of activity impacted by shortness of breath, mMRC results are divided into 0-4 grades. Grade 0 means no breathlessness except on strenuous exercise; grade 1 means shortness of breath when hurrying on the level or walking up a slight hill; grade 2 means walking slower than people of same age on the level because of breathlessness or having to stop to catch breath when walking at their own pace on the level; grade 3 means stoping for breath after walking ∼100 m or after few minutes on the level ground; and grade 4 means too breathless to leave the house, or breathless when dressing or undressing.
Change of chronic obstructive pulmonary disease Assessment Test (CAT) from baseline | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  The CAT is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. The CAT scale includes a total of 8 items, 0~5 points for each item. The total score ranges 0~40 points. Score of 0-10 points indicates slight impact; Score of 11-20 points indicates medium impact: Score of 21-30 points indicates serious impact; Score of 31-40 points indicates very serious impact.
Annual frequency of exacerbations | 1 year after treatment
  Frequency of exacerbations all through the year. A lower frequency means improvement of disease.
Symptoms, physical examination | Baseline, treatment day (D1), 24 hours after treatment, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal physical examination findings.
12-lead ECG | 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal 12-lead Electrocardiogram (ECG).
Blood routine | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal laboratory test results.
Urine routine | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal laboratory test results.
Blood biochemistry | Baseline, 4 weeks after treatment, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal laboratory test results.
Function of blood clotting | Baseline, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  Number of cases with abnormal function of blood clotting.
Carcinoembryonic antigen (CEA) | Baseline, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  CEA is a tumor marker used for early diagnosis of lung cancer.
Neuron-specific enolase (NSE) | Baseline, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  NSE is a tumor marker significantly elevated in small cell lung cancer.
Cytokeratin-19-fragment (CYFRA21-1) | Baseline, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  CYFRA21-1 is a tumor marker which is valuable for the pathological classification and prognosis evaluation of lung cancer.
Squamous cell carcinoma antigen (SCC) | Baseline, 12 weeks after treatment, 24 weeks after treatment, 52 weeks after treatment
  SCC is a specific marker for lung squamous cell carcinoma.Tumor markers are monitored to assess the safety.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of AMU, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No